CLINICAL TRIAL: NCT06197230
Title: The Effectiveness of Drawing Interventions on Depression Levels, Resourcefulness, and Spiritual Health of Older Adults in Nursing Homes
Brief Title: The Effectiveness of Drawing Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, IRNA KARTINA, Ms, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTUNHS_DI
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Older Adult
Keywords: Drawing Interventions; Depression; Resourcefulness; Spiritual Health; Older Adults
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized control trial with longitudinal design
Who Masked: Participant, Investigator
Masking Description: This intervention study is designed as single-blind; all the participants will be blinded to the allocation. To prevent participants from developing expectations regarding the intervention, they will be blinded to their group assignment.The investigator will not tell which is intervention and control group member
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group ; Drawing Intervention (Experimental): The intervention will be applied every week for 6 weeks. The level of depression, resourcefulness, spiritual resourcefulness, and spiritual health will be tested at the first week before the intervention (T0), the 3rd week (T1), the 6th week right after the interventions (T2), 1 month follow-up after the interventions (T3), and 2 months post-intervention.
  Interventions: Other: Drawing Intervention
- Control (Other): The control group will receive standard care in nursing home
  Interventions: Other: Drawing Intervention

INTERVENTIONS:
Other: Drawing Intervention — The primary sections of Drawing Intervention will be the "art-making" and "art-sharing" sections. During the art-making segment, the group leader will guide the participants through a paper-warming exercise before assigning them a specific subject to draw freely for 20-30 minutes. The leader will then ask participants to talk about the meaning of their artwork, encouraging them to explore their emotions regarding the theme and their drawing. This procedure will be implemented in each segment of the intervention (6 sessions).

SUMMARY:
The study will consist of two stages. The first stage of the study expects to find associations within dependent variables: depression level, resourcefulness, spiritual resourcefulness, and spiritual health in older adults. The second stage estimated that art drawing interventions will be effective for improving depression levels, resourcefulness, spiritual resourcefulness, and spiritual health.

DETAILED DESCRIPTION:
A cross-sectional research design will be used in the first stage, and the second stage of the research will be an intervention and longitudinal study with a randomized control trial design. In the first stage, four instruments will be applied, such as the Geriatric Depression Scale (GDS), Resourcefulness Scale (RS), Spiritual Resourcefulness Scale (SpRS), and Spiritual Screening Tool for Older Adults (SSTOA), to measure the levels of depression, resourcefulness, spiritual resourcefulness, and spiritual health of older adults at nursing homes in Indonesia. Three hundred older adults will be recruited through purposive sampling in the first stage of the study, while 128 participants will be recruited and randomized and assigned to both the experimental and control groups. There will be 64 subjects in each group. The art drawing intervention will be applied and last for 6 weeks in the experimental group. Five times of examinations about the related variables will be performed at the first week before intervention implemented (T0); the second measure will be performed 3 weeks after the intervention started (T1); 6 weeks of drawing intervention, the third examine will be tested (T2); and 1 and 2 months after the intervention completed, the participants will be asked to test for the T3 and T4

ELIGIBILITY:
Inclusion Criteria:

1. Currently live in nursing home
2. Have no physical impairment.
3. Have been staying in nursing home for at least 6 months.
4. Speak Bahasa Indonesia

Exclusion Criteria:

1. Have been diagnosed with psychiatric illness.
2. Have been diagnosed with severe physical disorders such as advanced cancer or motor impairments

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Geriatry Depression Scale (GDS) | 14 weeks
  Geriatric Depression Scale is one of depression scales known globally. The Geriatric Depression Scale (GDS), developed by Yesavage et al. in 1983, is a self-report instrument consisting of 30 items.
Resourcefulness Scale | 14 weeks
  The Resourcefulness Scale developed by Zauszniewski et al. (2006) will be used to test the degree of resourcefulness in older adults. The scale consists of 28-items on a 6-point Likert-type scale
Spiritual Health/Spiritual Self-assessment index for older adult | 14 weeks
  consists of 20 items, five measuring each of the constructs: (1) meaning and purpose, (2) hope and coping, (3) transcendence in relationships with God and others, and (4) religious practices. This tool offers options to the participants with a degree of agreement for each item using a five-point Likert scale. A numerical value will be assigned to each category: strongly disagree = 1, disagree = 2, uncertain = 3, agree = 4, and strongly agree = 5. Item responses total score that could range from 20 to 100. Higher scores indicated a greater degree of spiritual wellness. Each of the four subscales consisted of five items, permitting a scoring range from 5 to 25. Items one through five, representing measuring hope and coping; six through ten will measure transcendence; eleven through fifteen for meaning and purpose; and sixteen through twenty focused on religious practices.

CONTACTS AND LOCATIONS:
Overall Officials: Irna Kartina, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (2):
- Indonesia (2):
  - BPSTW Budi Luhur, Bantul, D.I Yogyakarta
  - Balai Pelayanan Sosial Tresna Wreda Unit Abiyoso, Yogyakarta, D.I Yogyakarta

IPD SHARING:
Plan to Share IPD: Undecided
Have not decided yet